CLINICAL TRIAL: NCT05202730
Title: Analgesic Effect of Peripheral Cutaneous Nerve Block of Knee Joint After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diwuweilong (Other)
Responsible Party: Sponsor-Investigator, Diwuweilong, Principal Investigator, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: KY20212115-F-2
Record Dates: First submitted 2021-12-05; First posted 2022-01-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Arthroplasty, Replacement, Knee; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional injection site and traditional local anesthetic formulation (Other)
  Interventions: Procedure: New local anesthesia injection site and new local anesthetic drug formulation.
- Traditional injection site and new local anesthetic formulation (Experimental)
  Interventions: Procedure: New local anesthesia injection site and new local anesthetic drug formulation.
- New injection site and traditional local anesthetic formulation (Experimental)
  Interventions: Procedure: New local anesthesia injection site and new local anesthetic drug formulation.
- New injection site and new local anesthetic formulation (Experimental)
  Interventions: Procedure: New local anesthesia injection site and new local anesthetic drug formulation.

INTERVENTIONS:
Procedure: New local anesthesia injection site and new local anesthetic drug formulation. — The traditional injection site is the posterior joint capsule and the popliteal artery space (iPACK) plus multiple layers of tissues around the knee joint (posterior joint capsule, ligaments and subcutaneous tissue). The traditional local anesthetic formulation is 1% ropivacaine 10ml+ normal saline 40ml+10mg Morphine + 5mg dexamethasone. The new local anesthesia injection site is iPACK+Knee Cutaneous Nerve Block. The new local anesthetic formula is 1% ropivacaine 10ml+ normal saline 40ml+10mg morphine+1ml triamcinolone acetonide.

SUMMARY:
Local anesthesia was performed on patients with total knee arthroplasty (TKA) through two different injection sites of local anesthetics and two local anesthetic drug . The pain score of patients after TKA was collected, then the analgesic effect of patients after TKA through two different injection sites and two different local anesthetic drug were analyzed and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients between the ages of 40-75, who meet the indications for total knee arthroplasty(TKA) surgery, plan to undergo unilateral TKA surgery, can tolerate surgical trauma, and have no surgical contraindications;
* 2. Patients who have good medical obedience and can cooperate to complete the evaluation of various indicators after the operation and continue to receive follow-up;
* 3. There is no contraindications to combined spinal-epidural anesthesia;
* 4. Agree to accept this trial and sign an informed consent form.

Exclusion Criteria:

* 1. Allergic to test drugs;
* 2. Abnormal liver, kidney or heart function;
* 3. People who have chronic pain symptoms in other parts of the body other than the knee joint;
* 4. Patients with a history of multiple operations on the knee joint, or patients with abnormal anatomical structures;
* 5. Patients who cannot perform early functional exercise after unconventional knee replacement or other systemic diseases;
* 6. Cannot communicate with researchers normally.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Change of the pain score before and after surgery | pre-operation, 6hours after surgery, 24hours after surgery, 48 hours after surgery.
  A Visual Analogue Scale (VAS) is used to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Xijing Hospital, The Air Force Medical University, Xi’an, Shanxi, China

REFERENCES:
- [Derived] Diwu W, Tang W, Yan M, Ma W, Xu H, Sun Q, Han Y, Wang Y, Wang C, Zhang D, Bi L, Yang M. Efficacy of Peripheral Cutaneous Nerve (PCN) on postoperative pain and functional outcome after total knee arthroplasty: a single-blind, randomized controlled clinical trial". BMC Anesthesiol. 2025 Jul 1;25(1):322. doi: 10.1186/s12871-025-03182-z. PMID 40597686